CLINICAL TRIAL: NCT00364780
Title: A Phase 2 Study of XL647 in Subjects With Non-Small-Cell Lung Cancer
Brief Title: Study of XL647 in Subjects With Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL647-201
Record Dates: First submitted 2006-08-14; First posted 2006-08-16 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — XL647

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients received XL647 at an intermittent dosing schedule receiving drug for 5 days followed by 9 days without drug.
  Interventions: Drug: XL647
- 2 (Experimental): Patients received drug at a daily dosing schedule
  Interventions: Drug: XL647

INTERVENTIONS:
Drug: XL647 — XL647 will be administered orally as a single agent. XL647 will be supplied as 50 mg tablets. Subjects in the Intermittent 5 & 9 cohort will receive XL647 at a dose of 350 mg on a 5 days on and 9 days off cycle every 2 weeks for 8 weeks. Subjects in the Daily Dosing cohort will receive XL647 administered daily as a single oral dose of 300 mg. In the absence of progressive disease (PD) and unacceptable XL647-related toxicity, subjects may continue to receive XL647 treatment on their assigned dosing schedule for up to 1 year on this study. Subjects who reach 1 year of treatment with no evidence of disease progression may, with the concurrence of the investigator and the sponsor, continue to receive therapy.

SUMMARY:
The purpose of this phase II study is to determine the safety, tolerability, and activity of XL647 in previously untreated subjects with non-small cell lung cancer (NSCLC). XL647 is a small molecule that potently inhibits multiple receptor kinases, including EGFR, VEGFR2 (KDR), ErbB2, and EphB4. Sensitivity to EGFR inhibitors has been linked to specific EGFR mutations and associated with certain clinical characteristics in patients with NSCLC (eg, female, minimal and remote smoking history, and adenocarcinoma histology).

ELIGIBILITY:
Inclusion Criteria:

* Subject has NSCLC with a histologically confirmed diagnosis of adenocarcinoma with measurable disease (stage IIIB, with malignant pleural effusion, and stage IV) and either has a demonstrated activating mutation of the EGF receptor in tumor tissue or meets one of three criteria: asian, female, and minimal or no smoking history.
* Measurable disease defined according to RECIST
* ECOG performance status of 0 or 1
* Normal organ and marrow function
* No other malignancies within 5 years, except for non-melanoma skin cancer

Exclusion Criteria:

* Radiation to ≥25% of bone marrow within 30 days of XL647 treatment
* Prior systemic anticancer therapy, including cytotoxic chemotherapy, anti-VEGF, anti-VEGFR, or anti-EGFR agents or investigational drug
* Subject has not recovered to ≤ grade 1 or to within 10% of baseline values from adverse events due to other medications administered > 30 days before study enrollment
* Receiving anticoagulation therapy with warfarin (low-dose warfarin < 1 mg/day, heparin and low molecular weight heparins are permitted)
* The subject meets any of the following cardiac criteria:

  * Corrected QT interval (QTc) of > 460 msec
  * Family history of congenital long QT syndrome or unexplained sudden death
  * History of sustained ventricular arrhythmias
  * Has a finding of left bundle branch block
  * Has an obligate pacemaker
  * Has important bradycardia defined as a heart rate of < 50 bpm due to sinus node dysfunction
  * Has uncontrolled hypertension
  * Has symptomatic congestive heart failure, unstable angina, or a myocardial infarction within the past 3 months
  * Has a serum potassium or serum magnesium level that falls outside the normal range
* The subject has progressive symptomatic or hemorrhagic brain or leptomeningeal metastases
* Uncontrolled intercurrent illness
* Subject is pregnant or breastfeeding
* Known HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-07; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Response rate | Inclusion until disease progression
Safety and tolerability | Inclusion until 30 days post last treatment

SECONDARY OUTCOMES:
Progression-free survival | Inclusion until disease progression or death
Duration of response | Inclusion until disease progression
Overall survival | Inclusion until 180-Day Follow-up post last treatment
Pharmacokinetic and pharmacodynamic parameters | At various time points from pre-dosing until post dosing

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - University of Chicago, Chicago, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wayne University, Wertz Clinical Cancer Center, Karmanos Center, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Case Western Reserve University, University Hospitals of Cleveland, Cleveland, Ohio

REFERENCES:
- [Background] Pietanza MC, Gadgeel SM, Dowlati A, Lynch TJ, Salgia R, Rowland KM Jr, Wertheim MS, Price KA, Riely GJ, Azzoli CG, Miller VA, Krug LM, Kris MG, Beumer JH, Tonda M, Mitchell B, Rizvi NA. Phase II study of the multitargeted tyrosine kinase inhibitor XL647 in patients with non-small-cell lung cancer. J Thorac Oncol. 2012 May;7(5):856-65. doi: 10.1097/JTO.0b013e31824c943f. PMID 22722787